CLINICAL TRIAL: NCT05907252
Title: The Effectiveness of Supervised Group-based Walking Program on Physical, Psychological and Social Outcomes Among Older Adults: A Randomized Controlled Trial
Brief Title: The Effectiveness of Supervised Group-based Walking Program Among Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HMRF05200108
Record Dates: First submitted 2023-05-02; First posted 2023-06-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Physical Inactivity; Social Interaction
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supervised Group-based Intervention (Experimental): Supervised Group-based intervention involves a professional walking fitness coach and 2 assistant coach. The coach is expected to require the participants to engage in the intervention in a form of group. The intervention groups will receive an 18-week walking training (3 sessions per week, 1 hour per session )in accordance with the intervention.
  Interventions: Behavioral: Supervised Group-based Intervention
- Non-supervised Group-based Intervention (Experimental): Supervised Group-based intervention involves no professional walking fitness coach; however, the research team member will ask the participants to engage in the intervention in a form of group, and complete the intervention according to goals and targets of each session. The intervention groups will receive an 18-week walking training (3 sessions per week, 1 hour per session )in accordance with the intervention.
  Interventions: Behavioral: Non-supervised Group-based Intervention
- Non-supervised Individual-based Intervention (Active Comparator): Non-supervised Individual-based Intervention involves no professional walking fitness coach; and no group forming is required. The participants will engage and complete the intervention individually. The intervention groups will receive an 18-week walking training (3 sessions per week, 1 hour per session )in accordance with the intervention.
  Interventions: Behavioral: Non-supervised Individual-based Intervention
- Control Group (No Intervention): Participants in the control group (CG) will not be arranged to participate in any walking or physical activity intervention during the whole study period (the 18-week intervention and 12-week follow-up periods), but they will be asked to keep a daily log on their physical activity, use of medicines, illness, and other health-related activities. Besides, the CG participants will be asked to report to the research resistant (RA) if a major change has been made in the aforementioned aspects. The RA will also check the daily logs of the participants through telephone or mobile phone every two weeks. Data from those who changed their normal lifestyles (especially taking up regular physical activity) will be excluded in the subsequent data analysis.

INTERVENTIONS:
Behavioral: Supervised Group-based Intervention — The intervention will be an 18-week walking program, with 3 times per week on alternative days. A 2-week basic walking practice with 3 sessions per week, 30-45 minutes per session, and being led by a certified walking trainer. The walking practice will take reference from the exercise procedure recommended by the "Healthy Exercise for All Campaign" (LCSD, Department of Health, and Physical Fitness Association Hong Kong, China, 2013). Upon completion of the 2-week basic walking practice, participants will enter week-3 to week-18 main walking program, in which the duration of each training session will increase to 45-70 minutes, depending on the levels of training. In the walking programs, the progressive training principle (ACSM, 2009) will be adopted, using 4 levels as prescribed, in which weeks 3 to 6 are Level-1; weeks 7 to 10 are Level-2, weeks 11 to 14 are Level-3, week 15-18 are Level-4.
  Arms: Supervised Group-based Intervention
Behavioral: Non-supervised Group-based Intervention — The intervention will be an 18-week walking program, with 3 times per week on alternative days. A 2-week basic walking practice with 3 sessions per week, 30-45 minutes per session, and without being led by a certified walking trainer. The walking practice will take reference from the exercise procedure recommended by the "Healthy Exercise for All Campaign" (LCSD, Department of Health, and Physical Fitness Association Hong Kong, China, 2013). Upon completion of the 2-week basic walking practice, participants will enter week-3 to week-18 main walking program, in which the duration of each training session will increase to 45-70 minutes, depending on the levels of training. In the walking programs, the progressive training principle (ACSM, 2009) will be adopted, using 4 levels as prescribed, in which weeks 3 to 6 are Level-1; weeks 7 to 10 are Level-2, weeks 11 to 14 are Level-3, week 15-18 are Level-4.
  Arms: Non-supervised Group-based Intervention
Behavioral: Non-supervised Individual-based Intervention — The intervention will be an 18-week walking program, with 3 times per week on alternative days. A 2-week basic walking practice with 3 sessions per week, 30-45 minutes per session, and without being led by a certified walking trainer. The walking practice will take reference from the exercise procedure recommended by the "Healthy Exercise for All Campaign" (LCSD, Department of Health, and Physical Fitness Association Hong Kong, China, 2013). Upon completion of the 2-week basic walking practice, participants will enter week-3 to week-18 main walking program, in which the duration of each training session will increase to 45-70 minutes, depending on the levels of training. In the walking programs, the progressive training principle (ACSM, 2009) will be adopted, using 4 levels as prescribed, in which weeks 3 to 6 are Level-1; weeks 7 to 10 are Level-2, weeks 11 to 14 are Level-3, week 15-18 are Level-4.
  Arms: Non-supervised Individual-based Intervention

SUMMARY:
Aim and Objectives:

The overall aim is to examine the effectiveness of supervised group-based walking intervention by comparing with non-supervised group-based walking and non-supervised individual-based walking interventions on improving physical, psychological and social outcomes among the older adults in Hong Kong. The outcomes of the research will be used as references for designing an effective walking operation manual for promoting healthy ageing among older adults in the community.

Objectives (Phase 1-Intervention):

1. To compare the differences of effects among supervised group-based, 5 non-supervised group-based, and non-supervised individual-based walking intervention programs, and the control group on the primary outcomes, including physical health, walking performance, loneliness, perceived social support and physical activity enjoyment among the older adults in Hong Kong.
2. To compare the differences of effects among supervised group-based, non-supervised group-based, and non-supervised individual-based walking intervention programs, and the control group on the secondary outcomes, including health-related quality of life and functional fitness among the older adults in Hong Kong.

(Please refer to Appendix D for the outcome measurements of the intervention) Objectives (Phase 2-Promotion)

1. To formulate and develop a walking operation manual for the use of implementing an effective walking program for the older adults in Hong Kong.
2. To promote and organize mass walking programs with the format as informed by the Phase 1 study among the older adults in the community (n=900-1080).
3. To raise the government's awareness towards the promotion of an effective walking program as informed by Phase 1 study for achieving the government's goal in promoting active aging.

DETAILED DESCRIPTION:
Justification for Conducting the Project:

(i) Health needs of the local community (supported by published data or relevant experiences) According to the World Health Organization, the number of people aged over 60 years old in the globe was increasing, while it has projected that this number will be increased by 40% in 2030 and by 110% by 2050. In Hong Kong, based on the statistics provided by the Office of Government Economist (2019), the proportion percentage growth of people aged 65 or above will almost be doubled in size to reach 31.9% in 2038.

Due to the reduced physical function and mobility caused by ageing, most of the older adults were highly committed to a sedentary lifestyle and being the most physically inactive population within a community. The research suggested that a longer duration of inactive or sedentary lifestyle could trigger various physical-related diseases and mental health problems, such as for overweight or obesity, diabetes, bone, and cardiovascular disorders, lower level of health-related quality of life, depression and loneliness. In particular, a longitudinal study in Hong Kong revealed that the physical and mental health of older adults were declining in the past 10 years. The study also indicated a reciprocal relationship between physical health and mental health, while mental health was shown to be the most interference factor due to the subsequent changes in physical health.

The lockdown and social restriction policy resulting from the prolonged COVID-19 pandemic has prevented older adults from going outdoors for exercise or social activities. This also worsened the level of physical activity, mental health, and subjective vitality. Research also showed that the degree of loneliness among older adults was significantly increased, as a result of the physical distancing, social isolation and worries about the COVID-19 pandemic.

To minimize the health consequences among older adults, physical activity is considered one of the most fundamental and effective forms of lifestyle interventions. The local studies revealed that physical activity was significantly associated with psychological well-being, including self-esteem, satisfaction and quality of life among Hong Kong older adults. Among various forms of physical activity, walking, which is with less restriction caused by the environment and equipment, hence, leading to better sustainability, is oneof the top choices of physical activity for older adults. Previous studies showed that regular walking could achieve better physical, functional and mental health among older adults, as well as lower mortality rate, facilitate weight loss, higher mobility, prevent chronic diseases and risk of falling, and generate positive psychological health, including vitality, independency, life satisfaction, subjective well-being and quality of life.

While WHO recommends adults to stay physically active, which means an accumulation of more than 150 minutes of moderate or above intensity or 75 minutes of vigorous-intensity of physical activity per week, it was found that only 36.5% of older adults in Hong Kong could meet the recommendation. An urgent effort to promoting a physically active lifestyle among our local older adults is needed, in which walking could be a better choice, especially for mass promotion.

(ii) Literature review on others' strategies to address these needs A recent systematic reviews and meta-analysis study concluded that nearly 43% of the research interventions on older adults were focused on strength, power and resistance training, 30% on mind-body exercises such as Tai Chi, Qigong and Yoga, while only 20% were on walking or mobility intervention. Although walking might be less popular than Tai Chi, walking was found to elicit almost 46% higher metabolic cost than Tai Chi, demonstrating as one of the most commonly recommended physical activities for older adults. Furthermore, walking is considered an essential component of outdoor mobility, it could be easily transformed into a transport model in order to replace driving or public transport. It was suggested that individuals should complete 8000 to 10000 steps per day for achieving better physical and mental health.

(iii) Scientific evidence supporting the strategies to address these needs proposed in this project Although walking is named as the most affordable type of physical activity for older adults due to the low risk of injury, as well as the likelihood of adopting and maintaining in daily life, walking-related research in Hong Kong, among older adults, in particular, is limited. For instance, two previous walking-related research studies in Hong Kong were focused on the prevention of falls and balance. Besides, there were only two walking-related research projects conducted under the Health and Medical Research Fund. Our research team had also conducted walking-related research among Hong Kong older adults from2014 to 2018, investigating the effects of residential physical and social environments on older adults' daily walking behaviours, as well as the walking habit among Hong Kong older adults. The results and findings of our walking studies have reaffirmed the needs of conducting an intervention study and promotion of walking for our local older adults.

Regarding the effectiveness of interventions, a systematic review and meta-analysis study stated that physical activity alone interventions showed inconsistent psychosocial outcomes, including social inclusion and loneliness, among older adults. Yet, a previous study reported that group-based physical activities showed greater contributions than individual-based physical activities on physical, psychological and social well-being among older adults. Subsequent studies on group-based intervention also showed improvement in social inclusion, loneliness and social interaction along with the social support structures involved in a group activity. Moreover, a meta-analysis study found that walking in a group could facilitate individuals' efficacy in walking thus significantly promote a higher level of physical activity. Similar results were also revealed in our research team's previous qualitative study (FRG2/17-18/009), suggesting that older adults would be better motivated in doing walking if they were assigned in a group and involved with social interaction. The research team's another research project also found better walking habit under companionships, social cohesion, encouragement and role models among the elderly participants (GRF Ref No.12620916). Furthermore, studies indicated that group-based physical activities with professional supervision showed benefits to older adults, especially in encouraging acceptable adaptations to perform various exercises or physical activities related to bones, muscles, and cardiovascular system, provided that physical activities can be performed whether in group-based or individual-based. A recent meta-analysis on older adults exercises interventions found that the findings from group exercise intervention trials were contradictory, in which further studies were encouraged to examine the disparities between groups and individual exercise intervention, as well as the impact of professional delivery and significant others on the results of exercise intervention.

When reviewing the walking-related programs in Hong Kong, the research team found that 2 local walking programs named as 'QualiWalk' (2013) and "Walk the City for Active Ageing" (2019). Both program implement a buddy-and-peer leader system by training young-olds as the program ambassador equipping them with knowledge of appropriate walking postures and leadership skills as well as aiming to assist walking groups for the older adults. Previous studies revealed that the buddy system with peer leadership could serve as a role model for the participants, thusproviding better connection and empathy towards individuals with similar age compared to a non-peer leader. The buddy system would a stronger motivation among the participants in adapting regular walking habits. However, the limitations of buddy system or peer leaders system were being less cost-effective and the researchers might found difficult to control the confounding factors created by the buddy/leader, such as the individual differences, the communication and management skills of the buddy in delivering the intervention. Hence, this might cause contrasting effects on promoting physical activity as well as on the outcomes of the intervention. Additionally, the 'QualiWalk' program did not provide regularly updated information and the effectiveness of the program was not clear to the public. Hence, it was difficult to reach those inactive older adults in the community, as well as failed to provide a scientific, documented, and sustainable walking program for the older adults in Hong Kong.

In order to advocate and achieve a Healthy Life Expectancy (HALE) in 2023, the World Health Organization recently released "Decade of Healthy Ageing Baseline Report" (WHO, 2020), aiming to promote healthy ageing through improving older adults' intrinsic capacity (both physical and mental capacities) and providing integrated care and services to respond to the needs of older adults. As referring to the integrated care and services mentioned in the WHO's report, it is believed that these services would less likely be achieved without involving professional guidance and social support environment. Also from the literature review, the previous studies have shown support to further studies adopting professional supervision and group-based intervention approaches. With the above significant references and recommendations, the research team has a strong justification for proposing the current study to examining whether a professionally supervised group-based walking program is more effective than non-supervised group-based as well as non-supervised individual-based walking programs on improving physical, psychological and social outcomes among the older adults in Hong Kong. The findings of this randomized controlled trial intervention study will shed light on the formats of the subsequent walking promotion program for the older adults in the community.

ELIGIBILITY:
Inclusion Criteria:

* Chinese older adults aged 65 years old or above
* capable of walking without assistive device
* healthy and living independently in communities
* being physically inactive

Exclusion Criteria:

* with cardiovascular or related diseases that prevent from intensive walking
* do not pass the PAR-Q screening or with physician's advice on the readiness of participation in walking training
* diagnosed with cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical Health Parameters - Body Composition | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Body Composition will be measured using the TANITA.
Physical Health - Resting Heart Rate | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Resting Heart Rate will be measured using the Fibit smart watch 2. Walking Performance The walking effects on participants' physical health parameters, including body composition, resting heart rate, and resting blood pressure will be assessed.
Physical Health - Resting Blood Pressure | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Both Systolic and Diastolic Resting Heart Rate will be measured. 2. Walking Performance The walking effects on participants' physical health parameters, including body composition, resting heart rate, and resting blood pressure will be assessed.
Walking Performance Walking Performance | During the procedure/intervention
  The time for completing the targeted steps in targeted heart rate zones of each participant in each training session will be recorded for analysis of performance and improvement on walking.
Psychological Outcomes - Loneliness | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Loneliness will be measured using the perceived loneliness scale.
Psychological Outcomes - Perceived social support | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Perceived social support will be measured using the Multidimensional Scale of Perceived Social Support Scale.
Psychological Outcomes - Physical Activity Enjoyment | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Physical Activity Enjoyment will be measured using the 8-item Physical Activity Enjoyment Scale (PACES).

SECONDARY OUTCOMES:
Health-related Quality of Life Score | Baseline Test: Before the intervention; Post-test:within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Health-related quality of life will be measured using the Short Form-36 (C-SF-36).
Functional fitness - Agility and dynamic balance | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Functional fitness Test based on the Senior Fitness Test (SFT) Manual.
Functional fitness - Lower Body Muscle Strength | Baseline Test: Before the intervention; Post-test: within 1 week after the intervention; Follow-up test: 3 months after the intervention (Assessing the change among the 3 time points)
  Functional fitness Test based on the Senior Fitness Test (SFT) Manual.

CONTACTS AND LOCATIONS:
Locations (1):
- Education University of Hong Kong, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Wong MYC, Leung KM, Thogersen-Ntoumani C, Ou K, Chung PK. Effectiveness of a supervised group-based walking program on physical, psychological and social outcomes among older adults: a randomised controlled trial protocol. BMJ Open. 2024 Oct 22;14(10):e088315. doi: 10.1136/bmjopen-2024-088315. PMID 39438105